CLINICAL TRIAL: NCT00199017
Title: Multicenter Trial for Treatment Optimization in T-lymphoblastic Lymphoma in Adults and Adolescents Older Than 15 Years (GMALL T-LBL 1/2004) (Amend 1)
Brief Title: German Multicenter Trial for the Treatment of Newly Diagnosed T-lymphoblastic Lymphoma in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMALL04
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2008-05

CONDITIONS: Lymphoma, Lymphoblastic
Keywords: T-LBL; Treatment; De novo; Chemotherapy; Adult; Lymphoma, lymphoblastic, T-cell
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma | interventions — Dexamethasone; Prednisolone; Cyclophosphamide; Vincristine; Daunorubicin; Asparaginase; Granulocyte Colony-Stimulating Factor; Mercaptopurine; Cytarabine; Methotrexate; Etoposide; Vindesine; Doxorubicin; Thioguanine; Cladribine

INTERVENTIONS:
Drug: Dexamethasone/Prednisolone
Drug: Cyclophosphamide
Drug: Vincristine
Drug: Daunorubicin
Drug: Asparaginase
Drug: G-CSF
Drug: Mercaptopurine
Drug: Cytarabine
Drug: Methotrexate
Drug: VP16
Drug: Vindesine
Drug: Adriamycin
Drug: Thioguanine
Drug: HDARAC
Procedure: CNS irradiation
Procedure: Mediastinal irradiation
Drug: Cladribine

SUMMARY:
This study evaluates the efficacy and tolerability of treatment for T-lymphoblastic lymphoma (T-LBL) according to a protocol for acute lymphoblastic leukemia. Patients receive one year of intensive cyclical chemotherapy with additional prophylaxis for central nervous system (CNS) relapse by intrathecal therapy and cranial irradiation and mediastinal irradiation after induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* T-lymphoblastic lymphoma (bone marrow [BM] involvement < 25%)
* Aged 15-65 years (55-65 years if biologically younger)
* Written informed consent

Exclusion Criteria:

* Severe complications due to lymphoma or secondary disease
* T-LBL as second malignancy or other active second malignancy
* Cytostatic pretreatment of LBL (exception of emergency treatments)
* Pregnancy
* Severe psychiatric illness or other circumstances which may compromise cooperation of the patient or informed consent
* Participation in other study interfering with study treatment

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2004-04; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
remission rate, remission duration, disease free survival, overall survival

SECONDARY OUTCOMES:
time and dose compliance, toxicity according to World Health Organization (WHO)

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD, PhD, Study Chair — University Hospital Frankfurt, Medical Dept. II
Locations (1):
- University Hospital, Medical Dept. II, Frankfurt, Germany

REFERENCES:
- See also: German Leukemia Trial Registry — http://www.studienregister-online.de